CLINICAL TRIAL: NCT06774469
Title: Effect of Overdose Ultrasound on the Articular Cartilage of the Osteoarthritic Knee in Adult Albino Rat: a Histological Study
Brief Title: Effect of Overdose Ultrasound on Osteoarthritic Knee in Adult Albino Rat: a Histological Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shahenda Mohamed Eissa, physiotherapist specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cu III F 89 23
Record Dates: First submitted 2024-12-24; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of Knee
Keywords: Osteoarthritis-ultrasound-overdose-albino rats-MIA-Articular cartilage
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections; Solutions; Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Masking Description: 40 rats
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- G1 (Control group) (Sham Comparator): (Normal group) For studying the normal histological structure of the articular knee joint. Will be assessed at the beginning of the study
  Interventions: Device: ultrasound
- G2 expermintal (Experimental): (Normal-US Group) Will be assessed after 30 consequent days
  Interventions: Device: assigned
- G3 expermintal (Experimental): (Osteoarthritis-induced group)Will be assessed after 14 days
  Interventions: Drug: Injection, Solution
- G4 expermintal (Experimental): (Osteoarthritis-Recovery group): Will be assessed after44 days
  Interventions: Drug: Injection, Solution
- G5 experimental (Experimental): (Osteoarthritis-US group) Will be assessed after 44 days
  Interventions: Device: assigned

INTERVENTIONS:
Device: assigned — Group II: (Normal-US Group): The rats will receive 2 sessions/ day of underwater pulsed US waves with 1 MHZ frequency and 1 watt/cm2 power, for 10 min for 30 consequent days applied to the right knee. The rats will be sacrificed after 30 days. Group V: (Osteoarthritis-US group) after two weeks of chemical induction of osteoarthritis, the rats will receive 2 sessions/ day of underwater pulsed US waves with 1 MHZ frequency and 1 watt/cm2 power for 10 min for 30 consequent days applied to the right knee. The rats will be sacrificed after 44 days.
  Arms: G2 expermintal; G5 experimental
Drug: Injection, Solution — Group III: (Osteoarthritis-induced group): For studying the histological changes of the articular knee joint after osteoarthritis induction in the right knee joint before recovery occur. The patellar ligament will be palpated below the patella and a single intra-articular injection of (MIA lateral to the ligament using an insulin syringe will be performed).
  The rats will be injected once with monosodium iodoacetate (MIA) dissolved in sterile saline (6 mg/kg body weight, 50 μL). Saline acts as a vehicle for MIA. The rats will be sacrificed after 14 days of MIA injection (1st day of the experiment).
  Group IV: (Osteoarthritis-Recovery group): The rats will be injected once with monosodium iodoacetate (MIA) dissolved in sterile saline (6 mg/kg body weight, 50 μL), Saline acts as a vehicle for MIA and will not receive any medication. The rats will be sacrificed after 44 days of MIA injection (1st day of the experiment).
  Other Names: MIA induction
  Arms: G3 expermintal; G4 expermintal
Device: ultrasound — Group I:Sham Comparator (Control group): for studying the normal histological structure of the articular knee joint.
  Arms: G1 (Control group)

SUMMARY:
The purpose of this study is to investigate the effect of overdose ultrasound on the articular cartilage of the osteoarthritic knee in adult albino rate. The US is considered the most popular and effective treatment for osteoarthritis as it can penetrate deep tissue reaching internal structures which allow it to be effective for osteoarthritis treatment. Previous researches apply US as a treatment for different cases with different intensity and repetition, but no one has actually proven the frequency of this use or the effect of excess use on cells, so the investigators need evidence to determine the optimum therapeutic dose and frequent repetition which should determine the effect of more than one session on the joint cartilage and cells and if it has a positive or negative effect and this is the main goal in this study which is limited in all studies concerning the US.

DETAILED DESCRIPTION:
Because many patients suffer from osteoarthritis and this work may help for treatment those patients. The US is considered the most popular and effective treatment for osteoarthritis as it can penetrate deep tissue reaching internal structures which allow to be effective for osteoarthritis treatment, also improves the cellular function by making microscopic gas bubbles near to the site of injury expand and contract rapidly, a process called cavitation. This process is thought to speed up the healing process in the injured body part. Previous researches apply US as a treatment for different cases with different intensity and repetition, but no one has actually proven the frequency of this use or the effect of excess use on cells, so the investigators need evidence to determine the optimum therapeutic dose and frequent repetition which should determine the effect of this repetition on the joints and cells and if has a positive or negative effect and this is the main goal in this study which is limited in all studies concerning the US in addition to previous systematic reviews regarding its effectiveness on KOA are outdated, and the latest reviews presented methodological limitations, such as the inclusion of mixed interventions, that hindered the evidence synthesis, and the inclusion of pulsed US (low-intensity) only.

The Investigators want to perform a more focused and comprehensive evidence synthesis targeting the isolated effects of the therapeutic US and specially the overdose to more clearly define its contributing role as an adjuvant treatment in rehabilitative regimens for KOA. Therefore studies worked on the effect of ultrasound on the knee cartilage especially femoral cartilage, the degradation and destruction of the femoral articular cartilage demonstrated a greater degree of deterioration than those of the tibial and patellar articular cartilage, and on some specific changes within its cells like apoptosis neglecting other cellular or matrix changes which may be affected by the destruction of articular cartilage and it's the second aim in this study. Although the results of previous studies suggest that US is a safe non-pharmacological treatment option that may provide additional pain relief and functional improvement in addition to cartilage repair with different parameters of US, no research assessing dosing regimen repetition to investigate its overdose effect on tissues and this was not reasonable to perform these analyses based on overdose on humans. This is the topic for the research, because the optimum therapeutic dose of therapeutic US is debated in previous research.

ELIGIBILITY:
Inclusion Criteria:

* Forty male Albino rats will be used for the study of knee osteoarthritis.
* At 7-8 weeks of age.
* 200-250 grams in weight will be obtained from the animal facility of the histology department, Faculty of Medicine, Tanta University.

Exclusion Criteria:

* Weight < 200-250 > kg.
* Rats with injured thighs and/or knees.
* Female rats.

Ages: 7 Weeks to 8 Weeks | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-03-09 (Estimated); Study Completion 2025-03-09 (Estimated)

PRIMARY OUTCOMES:
Samples to estimate the knee cartilage thickness (femoral cartilage) | at the begginig of the experiment and at the end
  captured by a microscope camera and analyzed using the Image J software (https://imagej.en.softonic.com) .
Samples to detect the morphology and the histological changes in cartilage matrix | at the begginig of the experiment and at the end
  Matrix changes can be detected by using different histochemical stains as a trichrome stain for the demonstration of collagen fibers and a combination of Van Gieson and Safranin O stains
Cellular changes | at the begginig of the experiment and at the end
  by studying and analyzing the hematoxylin and eosin stained section by using different lens powers of microscope.
Inflammatory changes | at the begginig of the experiment and at the end
  by immunohistochemical stains of CD markers according to the availability (either INOS or NF-KB).

CONTACTS AND LOCATIONS:
Overall Officials: Shereen Shawky Elabd, Assis. prof, Study Director — Tanta University
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt